CLINICAL TRIAL: NCT02457572
Title: Pulse Pressure Variation Measured During Valsalva Maneuver to Predict Fluid Responsiveness Under Open-chest Condition in the Patients Undergoing Off-pump Coronary Arterial Bypass Grafting
Brief Title: Pulse Pressure Variation Measured During Valsalva Maneuver to Predict Fluid Responsiveness Under Open-chest Condition
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hwan Lee, Assistant professor, Samsung Medical Center
Other Study IDs: SMC 2014-07-005
Record Dates: First submitted 2015-04-22; First posted 2015-05-29 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Cardiac Surgical Procedures; Thoracic Surgical Procedures; Sternotomy
MeSH Terms: interventions — Valsalva Maneuver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Valsalva maneuver: This is an observational study and as a diagnostic intervention, subjects in the study would receive valsalva maneuver. Valsalva maneuver was performed after sternotomy with the constant airway pressure of 30cmH2O for 2 breaths duration. The investigators perform this procedure to every patients and do not assign this intervention to the subjects of the study.
  Interventions: Procedure: Valsalva maneuver; Other: Fluid loading

INTERVENTIONS:
Procedure: Valsalva maneuver — Valsalva maneuver was performed after sternotomy with the constant airway pressure of 30cmH2O for 2 breaths duration.
  Other Names: Lung recruitment maneuver
Other: Fluid loading — We record the cardiac index values before and after volume expansion with 6ml/kg of balanced crystalloid
  Other Names: Balanced crystalloid infusion

SUMMARY:
Pulse pressure variation (PPV) is a well-known dynamic preload indicator to predict fluid responsiveness. However, its usefulness in open-chest conditions has been equivocal. The investigators evaluated whether PPV measured during Valsalva maneuver can predict fluid responsiveness after sternotomy.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients undergoing elective off-pump coronary arterial bypass grafting

Exclusion Criteria:

* Preoperative LV EF <= 35%
* Moderate or severe valvular heart disease
* Cardiac arrhythmia
* Intracardiac shunt
* Severe renal or liver disease
* Moderate to severe pulmonary hypertension (mean PAP > 35 mmHg)
* Patients with bullous lung disease or combined pneumothorax

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective off-pump coroanry arterial bypass grafting
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pulse pressure variation during Valsalva maneuver | during Valsalva maneuver

SECONDARY OUTCOMES:
Pulse pressure variation after sternotomy | 5 min after sternotomy

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Min JJ, Kim TK, Lee JH, Park J, Cho HS, Kim WS, Lee YT. Evaluation of augmented pulse pressure variation using the Valsalva manoeuvre as a predictor of fluid responsiveness under open-chest conditions: A prospective observational study. Eur J Anaesthesiol. 2017 May;34(5):254-261. doi: 10.1097/EJA.0000000000000613. PMID 28207430